CLINICAL TRIAL: NCT01455337
Title: Principal Investigator
Brief Title: Short-term Survival in Patients With Severe Alcoholic Hepatitis Treated With Steroid Versus Pentoxifylline
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Seung Ha Park, MD, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Alcoholic Hepatitis
Keywords: severe alcoholic hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Pentoxifylline; Prednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- prednisolone (Active Comparator)
  Interventions: Drug: Prednisolone
- pentoxifylline (Experimental)
  Interventions: Drug: pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline — 400mg tid
  Arms: pentoxifylline
Drug: Prednisolone — 40mg qd
  Arms: prednisolone

SUMMARY:
Alcoholic hepatitis represents one of the more serious forms of alcoholic liver disease. Critically ill patients with alcoholic hepatitis have high morbidity and mortality rate. Because of data suggesting that the pathogenic mechanisms in alcoholic hepatitis involve cytokine release and the perpetuation of injury by immunologic process, corticosteroid has been extensively evaluated in the treatment of alcoholic hepatitis. Although there are discrepancies in literature as several randomized trials and meta-analyses have reached contradictory results, corticosteroid for a subset of patients with severe alcoholic hepatitis, defined as a discriminant function ≥ 32, who also have no concomitant gastrointestinal bleeding, active infection, renal failure, and pancreatitis, has been recommended. This latter point emphasizes the important of meticulous selection to avoid the side effects of corticosteroid. Thus, the beneficial effects seems confined to a highly selected minority group in which the inhibitory effect of corticosteroid on liver inflammation is not outweighed by side effects such as weakened defense against infection, anti-anabolic effects, and possible ulcer-promoting effects causing gastrointestinal bleeding, which may be deleterious in these critically ill patients.

Newer understanding of the role of the role of TNF-α expression and receptor activity in alcoholic liver injury has prompted to an examination of TNF inhibition as an alternative to corticosteroid for severe alcoholic hepatitis. Pentoxifylline, a nonspecific TNF inhibitor, recently has been demonstrated in a randomized trial to improve survival in the therapy of severe alcoholic hepatitis. In particular, the survival benefit of pentoxifylline appears to be related to a significant reduction in development of hepatorenal syndrome. These results are promising, and support the need to further evaluate the potential of this new therapeutic avenue.

There is a need for head to head comparison of corticosteroid and pentoxifylline in severe alcoholic hepatitis. At the time the current study was designed (2008), corticosteroid was first-line treatment for severe alcoholic hepatitis. This study was designed to demonstrate that the effect of pentoxifylline was similar (i.e., not inferior) to that of prednisolone, an active form of prednisone. The aim of the present study was thus to compare the effects of pentoxifylline and prednisolone on the short-term mortality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Severe alcoholic hepatitis (discriminant function ≥ 32 points), Must be able to swallow tablets.

Exclusion Criteria:

* Gastrointestinal bleeding Bacterial infection HBsAg positivity Acute pancreatitis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
survival rate | at 1-month